CLINICAL TRIAL: NCT02353273
Title: The Pharmacokinetic Study of WH-1 Ointment in Subjects With Chronic Diabetic Foot Ulcers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Oneness Biotech Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ON101CLPK01
Record Dates: First submitted 2015-01-21; First posted 2015-02-02 (Estimated); Last update posted 2018-03-29 (Actual); Status verified 2018-03

CONDITIONS: Diabetic Foot
Keywords: WH-1,Diabetic Foot,Ulcer
MeSH Terms: conditions — Diabetic Foot

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- WH-1 ointment (Experimental): WH-1 ointment(1.25%),15g ointment per tube.
  Interventions: Drug: WH-1 ointment

INTERVENTIONS:
Drug: WH-1 ointment — Each subject will be applied the one dose of WH-1 ointment on Day 1, and twice a day of WH-1 application from Day 2 to Day 13, then one dose for Day 14.
  Other Names: No other intervention drug

SUMMARY:
The objective of this study is to evaluate the systemic exposures of WH-1 ointment which includes Salvigenin and Asiaticoside A in subjects with chronic diabetic foot ulcers following topical application of WH-1.

DETAILED DESCRIPTION:
This trial is designed as an open label, non-comparative study to evaluate the pharmacokinetic profiles of salvigenin and asiaticoside A in subjects who received the treatment of WH-1 ointment for diabetic foot ulcers. A total of 12 subjects will be completed in study. Each subject will be applied the one dose of WH-1 ointment on Day 1 following with the blood sampling collection, then twice a day of WH-1 application from Day 2 to Day 13, and another blood sampling collection scheduled on Day 14 after one dose application.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female is at least 20 years of age;
2. Diabetes mellitus (type I or II) was diagnosed with an HbA1c ≤ 12.0% measured during screening or within three months prior to randomization;
3. The target diabetic foot ulcer must have the following characteristics:

   1. ≤ Grade 2 per Wagner Ulcer Classification System;
   2. Lower limbs;
   3. No-infected;
   4. A cross-sectional area of between 1 and 25 cm2 post-debridement;
4. If female and of childbearing potential has a negative pregnancy test and is neither breastfeeding or intending to become pregnant during the study;
5. Able and willing to follow with study scheduled visits, comply with study procedures, and sign the informed consent.

Exclusion Criteria:

1. Acute Charcot' s neuroarthropathy as determined by clinical and/or radiographic examination;
2. Poor nutritional status defined as an albumin < 2.5 g/dL;
3. AST and/or ALT > 3X of the normal upper limit;
4. Clearance of Creatinine (Ccr) < 30 ml/min;
5. Treatment with immunosuppressive or chemotherapeutic agents, radiotherapy or systemic corticosteroids within 4 weeks prior to enroll;
6. A psychiatric condition (e.g., suicidal ideation), current or chronic alcohol or drug abuse problem, determined from the subject' s medical history, which, in the opinion of the Investigator, may pose a threat to subject compliance
7. Subjects who have received an experimental agent within 30 days, prior to enroll.
8. Subjects who have received WH-1 ointment within 30 days, prior to enroll.
9. Subjects who have history of smoking (define as more than 20 cigarettes per day) within 3 months prior to admission to the Hospital site.
10. Judged by the investigator not to be suitable for the study for any other reason.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2015-07-22 (Actual); Primary Completion 2016-07-05 (Actual); Study Completion 2016-09-05 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic parameters of Salvigenin and Asiaticoside A as listed below. (AUC0-∞, AUC0-t, Cmax)(Cmax,ss, AUC0-τ) | Day1; Day14
  AUC0-∞, AUC0-t, Cmax:
  1. Area under the concentration-time curve from time 0 to infinity (AUC0-∞)
  2. Area under the concentration-time curve from 0 to the time of last quantifiable level (AUC0-t)
  3. Maximum observed level (Cmax)
  Cmax,ss, AUC0-τ:
  1. Maximum observed plasma concentration at steady state (Cmax,ss)
  2. Area under the concentration versus time curve from time zero to the end of a dosing interval (AUC0-τ).

SECONDARY OUTCOMES:
Pharmacokinetic parameters of Salvigenin and Asiaticoside A as listed below, if appropriate. (Tmax, MRT, T1/2, Vd/F, CL/F) | Day1
  1. Time to peak concentration (Tmax)
  2. Mean residence time (MRT)
  3. Elimination half-life (T1/2)
  4. Apparent volume of distribution (Vd/F)
  5. Apparent clearance (CL/F)
Pharmacokinetic parameters of Salvigenin and Asiaticoside A as listed below, if appropriate. (Tmax,ss) | Day14
  Time to peak concentration at steady state (Tmax,ss)

CONTACTS AND LOCATIONS:
Overall Officials: Kai-Min Chu, Principal Investigator — Tri-Service General Hospital
Locations (1):
- Clinical Research Division, Taipei, Taiwan